CLINICAL TRIAL: NCT02533765
Title: Olaparib as Salvage Treatment for Cisplatin-resistant Germ Cell Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST186.02
Record Dates: First submitted 2015-06-17; First posted 2015-08-27 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Neoplasms, Germ Cell and Embryonal
Keywords: Cisplatin-resistant; Neoplasms, Germ Cell and Embryonal; Salvage treatment; olaparib
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olaparib (Experimental): Olaparib 300mg twice daily continuously
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib dispensed to patients at the dose of 300 mg twice daily (BID) continuously until the patient completes the study, withdraws from the study or closure of the study.
  Other Names: AZD2281

SUMMARY:
This is open-label, single-arm, two-stage phase II trial of olaparib in patients with relapsed/refractory metastatic germ cell cancer. The primary objective is to evaluate the preliminary activity of Olaparib in GCT tumors. The secondary objective is to evaluate the safety of Olaparib in patients with cisplatin-refractory GCT.

DETAILED DESCRIPTION:
This is a proof-of principle open-label, single-arm, two-stage phase II trial of olaparib 300 mg twice daily in patients with relapsed/refractory metastatic germ cell cancer. The study will recruit 10 patients, if no response is seen the study is terminated. If one or more responses are observed, further 19 patients (for a total of 29 patients) will be enrolled. If 4 or more of the first 29 evaluable patients have achieved objective response, further studies in patients with metastatic germ cell cancer are warranted.

The main inclusion criteria are:

* Patient with metastatic gonadal GCT or extragonadal GCT originating from retroperitoneum or mediastinum.
* Disease progression during cisplatin-based chemotherapy or disease progression or relapse after high-dose chemotherapy or disease progression or relapse after at least 2 different cisplatin-based regimens
* At least one measurable lesion that can be accurately assessed by CT/MRI/plain x-ray) at baseline and follow up visits.

The study will be analyzed on an intent-to-treat basis. Secondary parameters will be analyzed exploratively for the intent-to-treat population.

Correlations between with biomarkers (PAR, poly adenosine diphosphate-ribose polymerase (PARP-1), PTEN, XPA, ERCC1-3, XPF, FanD2, γ-H2AX) expression in paraffin-embedded tumor samples and clinical outcome will be performed in an exploratory intent. Plasma samples will be collected at baseline and at response/progression for possible retrospective biomarkers study.

ELIGIBILITY:
Inclusion criteria:

1. Patients ≥ 18 years old
2. Histologically verified metastatic gonadal GCT or extragonadal GCT originating from retroperitoneum or mediastinum.
3. Disease progression during cisplatin-based chemotherapy or disease progression or relapse after high-dose chemotherapy or disease progression or relapse after at least 2 different cisplatin-based regimens
4. patients who progressed during cisplatin-based therapy and who are not eligible for high-dose chemotherapy
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0-2
6. Life expectancy ≥3 months
7. At baseline adequate function of liver, kidneys and bone marrow

   * Neutrophils ≥ 1500 /mm3;
   * Hemoglobin ≥ 9.0 g/dL;
   * Platelets ≥ 80 x109/L;
   * Creatinine ≤ 1.5x upper limit of normal (ULN) In case of liver metastases increased levels of the following three parameters is acceptable:
   * Bilirubin ≤ 1.5 x ULN
   * serum glutamate oxaloacetate transaminase (SGOT (AST) ≤2.5 x ULN
   * serum glutamate pyruvate transaminase (SGPT (ALT) < 2.5 x ULN;
8. Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Conference on Harmonization Good Clinical Practice (ICH GCP), and national/local regulations.Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
9. At least one measurable lesion that can be accurately assessed by CT/MRI/plain x-ray) at baseline and follow up visits.

Exclusion criteria:

1. Systemic antitumor treatment within 21 days before study entry
2. Simultaneous radiotherapy to the only target lesion
3. Patients with resting ECG with QTc > 470 msec detected on 2 or more time points within a 24 hour period or family history of long QT syndrome. If ECG demonstrates QTc >470 msec, patient will be eligible only if repeat ECG demonstrates QTc ≤470 msec
4. Patients who have experienced a seizure or seizures within 6 months of study treatment or who are currently being treated with cytochrome P450 enzyme inducing anti-epileptic drugs for seizures.
5. Patients with uncontrolled brain metastases.
6. Patients receiving prohibited classes of inhibitors of CYP3A4 (see section 6.5.1).
7. Patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
8. Patients with any acute toxicities due to previous cancer treatment that have not resolved to a Common Toxicity Criteria for Adverse Effects (NCI-CTCAE v 4.03) grade 0 or 1 with the exception of chemotherapy induced alopecia and grade 2 peripheral neuropathy.
9. Patients affected by myelodysplastic syndrome or acute myeloid leukemia
10. Known to be serologically positive for HIV and receiving antiretroviral therapy
11. Known seropositive for active viral infection with hepatitis B virus (HBV) (patients who are HBsAg negative, anti-HBs positive and/or hepatitis B core antigen (Anti-HBc) positive, but viral DNA negative are eligible)
12. Known seropositive for active infection with hepatitis C virus (HCV)
13. Patients unwilling or unable to comply with the protocol
14. Patients with unstable angina pectoris, myocardial infarction ≤ 6 months prior to first study treatment, congestive heart failure New York Heart Association (NYHA) III-IV or serious uncontrolled cardiac arrhythmias
15. Patients with an active or uncontrolled infection
16. Patients who have a history of another primary malignancy and are off treatment for ≤ 3 years, with the exception of non-melanoma skin cancer
17. Patients who have undergone major surgery within 4 weeks prior to starting study drug (e.g. intra-thoracic, intra-abdominal, or intra-pelvic) or significant traumatic injury, or who have not recovered from the side effects of any of the above within 6 weeks
18. Patients who have participated in another interventional clinical trial within 30 days before study entry
19. Other serious medical conditions that could impair the ability of the patient to participate in the study
20. Active infection requiring systemic antibiotic-, anti-viral-, or anti-fungal medication
21. Active cancer (other than GCT) including prior malignancy from which the patient has been disease-free for ≤3 years (except superficial basal cell skin cancer)
22. Patients with a known hypersensitivity to the combination/comparator agent
23. Patients with uncontrolled seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 30 months
  The percentage of patients whose cancer achieve either a partial response or a complete response.Tumor response will be assessed using CT scan or MRI of chest/abdomen using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and by tumor marker (AFP, betaHCG, LDH) measurements

SECONDARY OUTCOMES:
Evaluation of number, type and grade of Adverse Events | Up to 30 months
  All patients will be evaluable for toxicity from the time of their first treatment with Olaparib
Progression free survival (PFS) | Up to 30 months
  time from the date of starting of the treatment to the date of the first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
Overall survival (OS) | Up to 30 months
  Time from enrolment to the date of death due to any cause. For subjects with no known date of death, survival time will be censored at the date of their last on-study assessment.
exploratory analysis of the association between PFS or OS and biomarkers | Up to 30 months
  correlation between biomarkers (PAR, PARP-1, PTEN, XPA, ERCC1-3, XPF, FanD2, γ-H2AX) in paraffin-embedded tumor samples and plasma with clinical outcome (response, PFS, OS)

CONTACTS AND LOCATIONS:
Overall Officials: Ugo De Giorgi, MD, Principal Investigator — IRST IRCCS, Meldola; Sandro Pignata, MD, Principal Investigator — Istituto Nazionale Tumori di Napoli
Locations (2):
- Italy (2):
  - U.O Oncologia Medica, IRST IRCCS, Meldola, FC
  - Istituto Nazionale Tumori IRCCS "Fondazione G.Pascale", Napoli